CLINICAL TRIAL: NCT01952639
Title: Postprandial Muscle Protein Synthesis Following Wheat Protein Ingestion in Vivo in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Stefan Gorissen, MSc, Maastricht University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: METC 13-3-045; NL45958.068.13 (Registry Identifier: Dossiernummer CCMO)
Record Dates: First submitted 2013-09-23; First posted 2013-09-30 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 30 g of wheat protein (Experimental): Subjects will consume 30 g of wheat protein protein type and amount
  Interventions: Dietary Supplement: protein type and amount
- 30 g of wheat protein hydrolysate (Experimental): Subjects will consume 30 g of wheat protein hydrolysate protein type and amount
  Interventions: Dietary Supplement: protein type and amount
- 30 g of whey protein (Active Comparator): Subjects will consume 30 g of whey protein protein type and amount
  Interventions: Dietary Supplement: protein type and amount
- 30 g of casein (Active Comparator): Subjects will consume 30 g of casein protein type and amount
  Interventions: Dietary Supplement: protein type and amount
- 60 g of wheat protein hydrolysate (Experimental): Subjects will consume 60 g of wheat protein hydrolysate protein type and amount
  Interventions: Dietary Supplement: protein type and amount

INTERVENTIONS:
Dietary Supplement: protein type and amount — Subjects will stay in a supine position and consume a test beverage containing different amounts ans types of protein

SUMMARY:
Rationale: The progressive loss of skeletal muscle mass with aging, or sarcopenia, has a major impact on our health care system due to increased morbidity and greater need for hospitalization and/or institutionalization. One way to prevent skeletal muscle loss is to improve dietary intake of the elderly. Both whey and casein seem to offer an anabolic advantage over soy protein for promoting muscle hypertrophy. As a consequence it is assumed that (all) plant based proteins have less potent anabolic properties when compared with animal based proteins. However, there is little theoretical background for such assumptions.

Objective: To provide evidence for the efficacy of wheat protein and wheat protein hydrolysate when compared with milk proteins (i.e. whey and casein) as a dietary protein to stimulate postprandial muscle protein synthesis in vivo in healthy older humans.

Study design: double-blind, placebo-controlled intervention study Study population: 60 healthy non-obese (BMI 18.5-30 kg/m2) older males (age: 65-80 y) Intervention: A protein beverage (350 mL) containing 30 g of whey, casein, wheat protein, or wheat protein hydrolysate or 60 g of wheat protein hydrolysate will be consumed (n=12 per group).

Main study parameters/endpoints: Primary study parameters include muscle protein synthesis rates. Secondary study parameters include whole-body protein synthesis, breakdown, oxidation, and net balance.

Hypotheses: We hypothesize that ingestion of wheat protein hydrolysate results in a greater muscle protein synthetic response when compared with the intact wheat protein due to its faster digestion and absorption. Furthermore, ingestion of wheat protein hydrolysate results in a higher muscle protein synthetic response when compared with casein, but lower when compared with whey protein. Ingestion of 60 g of wheat protein hydrolysate (amount of leucine equal to 30 g of whey protein) will result in a similar muscle protein synthetic response compared to ingestion of 30 g of whey protein.

DETAILED DESCRIPTION:
Aging is accompanied by a progressive decline in skeletal muscle mass. This age-related loss of muscle mass, or sarcopenia, is attributed to an imbalance between muscle protein synthesis and breakdown. As basal muscle protein synthesis rates do not seem to differ between young and elderly, most research has focused on potential impairments in the muscle protein synthetic response to the main anabolic stimuli, i.e. food intake and exercise. Skeletal muscle protein synthesis is highly responsive to food intake in healthy young adults. Recent data indicate that the muscle protein synthetic response to food intake may be blunted in the elderly. This proposed anabolic resistance is now being regarded as a key factor in the etiology of sarcopenia. Effective strategies to prevent and/or counteract the age-related loss of muscle mass include protein supplementation, preferably in combination with resistance exercise. Recent studies show the efficacy of dietary protein supplementation to improve muscle strength and function in frail elderly and to further augment the gains in muscle mass and function when combined with resistance exercise. As a consequence, nutrition research is now looking for the optimal amount, type, and timing of protein consumption to maximize postprandial muscle protein synthesis rates.

Improvements in protein balance and/or higher muscle protein synthesis rates have been reported following the ingestion of various types of dietary protein: whey, casein, soy, casein hydrolysate, egg protein, and whole-milk and/or fat-free milk. It seems obvious to question which source of dietary protein is most effective in promoting muscle protein synthesis. There is only limited research comparing the efficacy of the ingestion of different proteins sources on the protein synthetic response. As such, it is difficult to identify a specific protein source that is most potentiating. This is further complicated by the fact that numerous parameters modulate the muscle protein synthetic response to protein ingestion. The amount and timing of protein administration, the amino acid composition of the protein, and the digestion and absorption kinetics of the protein source (or mixed meal), may all modulate the muscle protein synthetic response.

Milk proteins, i.e. whey and casein, are the most widely studied dietary proteins. Casein and whey seem to have distinct anabolic properties, which are attributed to differences in digestion and absorption kinetics. Whey protein is a soluble protein that leads to fast intestinal absorption, whereas intact casein clots in the stomach delaying its digestion and absorption and the subsequent release of amino acids in the circulation. The faster, but more transient rise in plasma amino acid concentration after whey protein ingestion can lead to higher protein synthesis rates. In addition to intrinsic differences in digestion and absorption rate, it has been suggested that whey protein can more effectively stimulate protein synthesis due to its greater leucine content when compared to casein. Both whey and casein seem to offer an anabolic advantage over soy protein for promoting muscle hypertrophy. As a consequence it is assumed that (all) plant based proteins have less potent anabolic properties when compared with animal based proteins. However, there is little theoretical background for such assumptions. In this study we will assess the capacity of wheat protein ingestion as a means to increase postprandial muscle protein synthesis in vivo in humans. By directly comparing the anabolic properties of wheat protein or wheat protein hydrolysate with both casein and whey, we will determine the anabolic properties of wheat protein (hydrolysate) in vivo in older humans.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males
* Age between 65 and 80 y
* BMI between 18.5 and 30 kg/m2

Exclusion Criteria:

* Wheat allergy
* Celiac disease
* Lactose intolerance
* Smoking
* Diabetes
* Diagnosed GI tract diseases
* Arthritic conditions
* A history of neuromuscular problems
* Any medications known to affect protein metabolism (i.e. corticosteroids, non-steroidal anti-inflammatories, or prescription strength acne medications).
* Use of anticoagulants
* Participation in exercise program
* Hypertension, high blood pressure that is above 140/90 mmHg.

Ages: 65 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
muscle protein synthesis (MPS) rates | Change in MPS from baseline after ingestion of different types of protein (baseline vs. postprandial period (0-5h))

SECONDARY OUTCOMES:
whole-body protein metabolism | Change in whole-body protein metabolism from baseline after ingestion of different types of protein (baseline vs. postprandial period (0-5h))
  Whole-body protein metabolism consists of protein breakdown, synthesis, oxidation, and net balance. This will assessed by measuring plasma enrichments of the infused and ingested tracers and calculate the endogenous rate of appearance (breakdown), total rate of disappearance (synthesis), oxidation, and net protein balance (synthesis - breakdown).

CONTACTS AND LOCATIONS:
Overall Officials: Luc JC van Loon, Prof. Dr., Principal Investigator — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

REFERENCES:
- [Derived] Gorissen SH, Horstman AM, Franssen R, Crombag JJ, Langer H, Bierau J, Respondek F, van Loon LJ. Ingestion of Wheat Protein Increases In Vivo Muscle Protein Synthesis Rates in Healthy Older Men in a Randomized Trial. J Nutr. 2016 Sep;146(9):1651-9. doi: 10.3945/jn.116.231340. Epub 2016 Jul 20. PMID 27440260